CLINICAL TRIAL: NCT05492617
Title: Early Detection of de Novo Cancer in Liver Transplant Recipients - a ScandiaTransplant Collaboration
Brief Title: Early Detection of de Novo Cancer in Liver Transplant Recipients
Acronym: DETECT
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Hans-Christian Pommergaard, MD, PhD, Associate Professor, Rigshospitalet, Denmark
Other Study IDs: The DETECT study
Record Dates: First submitted 2022-08-05; First posted 2022-08-08 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: De Novo Cancer; Liver Transplant Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background The risk of cancer in liver transplant recipients is twice the cancer risk in the general population and de novo cancers are one of the leading causes of death after liver transplantation. The immunosuppressive medication, used to prevent organ rejection, is considered a key factor increasing the risk of de novo cancer.

Objectives I. Determine prevalence and incidence of de novo cancer in liver transplant recipients and build an algorithm to identify high-risk individuals II. Investigate if opportunistic viral infections (as a surrogate for over-immunosuppression) is associated with non-virus associated de novo cancers III. Investigate if cell free DNA fragmentation can be used to identify liver transplant recipients with de novo cancers and to identify cancer at an asymptomatic stage

Methods The study is in collaboration with all five Scandinavian liver transplant centers in ScandiaTransplant (Copenhagen, Oslo, Gothenburg, Stockholm and Helsinki) and includes all liver transplant recipients from the centers. Data on demographics, de novo cancer and risk factors are retrieved from electronic health records, cancer registries and the ScandiaTransplant database (n=3628). Blood samples to perform viral and cell free DNA fragmentation analyses are retrieved from the biobank at Rigshospitalet (n=932).

Implications The study includes a large cohort of liver transplant recipients from all of Scandinavia. With cancer as one of the primary causes of death in liver transplant recipients, new tools are needed to identify recipients with increased risk of developing de novo cancer. In particular, new tools allowing early diagnosis of de novo cancer enabling curative intended intervention. The study has potential to identify liver transplant recipients with increased risk of developing de novo cancer and reduce cancer related mortality.

DETAILED DESCRIPTION:
BACKGROUND Liver transplantation is a complex surgical procedure and the only curative treatment for many patients with chronic end-stage liver disease and acute liver failure. Short-term survival for liver transplant recipients has improved markedly over the past decades with a 1-year survival of 90%[1]. In contrast, over the same time period there has been no improvement in long-term survival, with only 61-74% of liver transplant recipients living 10 years after transplantation [2, 3]. This is despite the median age at time of transplantation being 48 years. De novo cancer after transplantation is one of the leading causes of late death and an independent risk factor for mortality after liver transplantation [3, 4].

The cumulative incidence of de novo cancer after liver transplantation in the Scandinavian population is 1% at 1 year, 3% at 3 years, 4% at 5 years, 9% at 10 years, and 15% at 20 years [5]. Risk of de novo cancer for liver transplant recipients is twice the cancer risk in the general population [5, 6] and even higher for children and adolescents [3]. In addition, cancers present at a more advanced stage [6]. After liver transplantation lifelong immunosuppressive treatment is necessary to prevent organ rejection. Immunosuppression is considered as a primary risk factor for de novo cancer [7-10], likely due to impaired cancer surveillance [8].

While there are no reliable biomarkers reflecting the status of the immune function in liver transplant recipients, opportunistic infections with Cytomegalovirus (CMV) and Torque Teno Virus (TTV), have shown to act as surrogate measures for over-immunosuppression. In contrast to Epstein-Barr virus (EBV) and human herpes virus 8 (HHV8), CMV and TTV have not been directly implicated in the pathogenesis leading to cancer and these viruses may therefore serve as functional markers for the level of immunosuppression [11-13]. The relationship between opportunistic virus infections and non-virus associated de novo cancers after liver transplantation has not been sufficiently investigated.

Due to high incidence of cancer, screening may be relevant in liver transplant recipients [14, 15]. Positron Emission Tomography-Computed Tomography (PET-CT) is the method of choice to detect de novo cancers, but the modality is costly and carries a risk of false positive results [16]. The method genome-wide cell free DNA fragmentation allows differentiation between cell free DNA from healthy individuals and patients with cancer [17]. In a previous study, early detection of various cancers was possible with a high accuracy (area under curve (AUC) of 0.94). Moreover, tissue of origin could be identified from fragmentation profiles. This method has not been investigated in liver transplant recipient and may be used to screen recipients, who could benefit from further investigations such as PET-CT.

In conclusion, to reduce cancer related mortality in liver transplant recipients, new tools are needed to identify recipients with increased risk of developing de novo cancer. In particular, new tools are needed that will allow diagnosis of de novo cancer at an early time-point that allows curative intended intervention. The study has potential to provide information to close important gaps in our knowledge and to improve the prognosis in liver transplant recipients.

OBJECTIVES

The overall objectives of the present study is to reduce de novo cancer mortality in liver transplant recipients. To obtain this goal, we will:

I. Determine prevalence and incidence of de novo cancer in liver transplant recipients in Scandinavia and build an algorithm to identify high-risk individuals II. Investigate if opportunistic viral infections (as a surrogate for over-immunosuppression) is associated with the non-virus associated de novo cancers III. Investigate if cell free DNA fragmentation can be used to identify liver transplant recipients with de novo cancers, and to identify cancer at an asymptomatic stage

METHODS This study is a multicenter cross-sectional case-control study in liver transplant recipients, aged between 20 and 100 years, from five Scandinavian liver transplantation centers (Copenhagen, Oslo, Gothenburg, Stockholm, Helsinki). These centers collaborate in the organ exchange organization Scandiatransplant with the aim to promote research and develop organ donation, allocation and transplantation. The past decade 3628 liver transplant recipients have been registered in the Scandiatransplant database, and all will be included in the study [18, 19, 20].

Plasma, serum and whole blood samples, collected pre-liver transplantation and sequentially during post-liver transplantation follow-up, from recipients in Scandinavia has been stored in a dedicated biobank at Rigshospitalet (n=932). Inclusion is ongoing and we expect to have included additionally 300 patients at the time of the proposed analyses.

From local cancer registries, cancer type and date of diagnosis will be registered, and from the Scandiatransplant database and electronic records, clinical variables will be retrieved. These include age, gender, immunosuppressive regime and duration incl. tacrolimus levels, acute rejections, liver biopsy findings, indication for liver transplantation, alcohol and smoking history, and co-morbidity.

CMV & TTV In a nested case-control study among 67 liver transplant recipients with cancer and 207 liver transplant recipients without cancer, blood samples are investigated for TTV-DNA and CMV-DNA as independent risk faktors for cancer after liver transplantation. Previous studies have shown TTV viral load to be associated with the intensity of immunosuppression [11, 13], why TTV viral load can be used as a marker of immunosuppression. Although more than 80% of adults are CMV-seropositive, detectable CMV viral replication is less common. For CMV, we will use detectable CMV replication as a marker of over-immunosuppression [12, 21]. Detection and quantification of CMV-DNA in blood is performed as a routine analysis at the Department of Clinical Microbiology, Rigshospitalet under CE-IVD on the Roche cobas 6800-platform and is quality assured externally and calibrated according to WHO's international standard. For the detection and quantification of TTV-DNA, the Biomerieux Argene TTV R-GENE assay is used: DNA is purified on Qiagen Qiacube and real-time PCR is performed on Agilent AriaMx. Measurement of TTV-DNA is performed as research only, as the analysis has not yet been established as routine operation. Nikolai Kirkby is responsible for the execution and quality assurance of the analyzes for CMV / TTV-DNA.

Cell-free DNA Fragmentation In a case-control study, blood samples from the biobank are examined with cell-free DNA fragmentation among 67 liver transplant recipients with cancer and 207 matched controls. Cell-free DNA in plasma is analyzed by shallow whole genome sequencing and DELFI (DNA evaluation of fragments for early interception). DELFI is a machine learning algorithm developed by members of the project group. It is used to detect cancer and the tissue the cancer originates from by examining fragment size and pattern of cell-free DNA [17]. In recipients where a cancersignal is measured, blood samples prior to the cancer diagnose will be analyzed to investigate if the method is able to detect cancer prior to clinical symptoms. Cell-free DNA fragmentation analyzes are performed at the Department of Molecular Medicine, University of Aarhus by Claus Lindberg Andersen.

STATISTICS The prevalence and incidence of de novo cancer in liver transplant recipients is determined. To asses risk factors, Cox multivariate regression analysis is applied with time to first de novo cancer diagnosis after liver transplantation as a dependent variable.

To establish an algorithm reflecting the risk of de novo cancer after liver transplantation, hazard ratios (HR) from significant variables in the multivariate COX-regression will be transformed with natural logarithm to enable addition. The score will be expressed by the exponential function of this summation (i.e. exp [ln (HR 1) + ln (HR 2) + ln (HR n)]).

We will compare the standard deviations from cell free DNA fragmentation profiles between cases and controls by a Wilcoxon rank sum test.

POWER In liver transplant recipients, TTV viremia at three months after liver transplantation increased with increasing immunosuppression [13]. Viremia increased from 5.8 log10 copies/ml in low dose monotherapy immunosuppression to 7.3 log10 copies/ml in combination treatment. Given an alpha of 0.05 and a power of 0.90 with 67 cases and 201 control, the minimal detectable difference in TTV viremia will be 0.4 log10 copies/ml (G*Power, version 3.1.9.3).

In a previous study, 73% of cancer cases were identified with DELFI and cancer signal was only seen in 1.9% of healthy controls [17]. However, cancer patients and healthy control may not be comparable to liver transplant recipients with respect to DELFI analyses. Due to risk of inflammation/rejection, we suspect a higher risk of a cancer signal in the control group. Given an alpha of 0.05 and a power of 0.90 with 67 cases and 201 controls, the minimal detectable difference in proportion will be 21% (73% in cases and 52% in controls) (G*Power, version 3.1.9.3). Median time from blood sampling to freezing for our plasma samples is less than 3 hours, which is acceptable for cell free DNA fragmentation analyses.

ELIGIBILITY:
Inclusion Criteria:

* All liver transplant recipients from the five centers between 20 and 100 years of age at time of transplantation, during the period 1.1.2010 - 31.12.2020 are included in the study (n=3628)
* For the nested case-control study: Plasma, serum and whole blood samples, collected pre-liver transplantation and sequentially during post-liver transplantation follow-up, from recipients in Scandinavia has been stored in a dedicated biobank at Rigshospitalet (n=932). Inclusion is ongoing and we expect to have included additionally 300 patients at the time of the proposed analyses.

Exclusion Criteria:

* Cancers arisen first 30 days post liver transplantation are excluded as it is considered a to be delayed diagnosis of pre-liver transplantation and not a de novo cancer.
* Donor-derived cancers or a relapse or metastatic disease from a cancer diagnosed prior to liver transplantation are excluded.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is a multicenter cross-sectional case-control study in liver transplant recipients, aged between 20 and 100 years, from five Scandinavian liver transplantation centers (Copenhagen, Oslo, Gothenburg, Stockholm, Helsinki). These centers collaborate in the organ exchange organization Scandiatransplant with the aim to promote research and develop organ donation, allocation and transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 3628 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence and Prevalence of De Novo Cancer in Liver Transplant Recipients | 2010-2020
  Solid and hematological cancers according to the ICD-11.
CMV & TTV association with De Novo Cancer in Liver Transplant Recipients | 2010-2020
  We will investigate if detectable/higher levels of CMV- and TTV is predictive of the development of de novo cancer in liver transplant recipients through a nested case-control study.
Cell-free DNA fragmentation to identify liver transplant recipients with de novo cancer at an asymptomotic stage | 2010-2020
  Cell-free DNA in plasma is analyzed by shallow whole genome sequencing and DELFI (DNA evaluation of fragments for early interception). DELFI is a machine learning algorithm developed by members of the project group. It is used to detect cancer and the tissue the cancer originates from by examining fragment size and pattern of cell-free DNA.
  The study is designed as a nested case-control study.